CLINICAL TRIAL: NCT03594747
Title: A Phase 3, Multicenter, Randomized Open-Label Study to Compare the Efficacy and Safety of Tislelizumab (BGB A317, Anti-PD1 Antibody) Combined With Paclitaxel Plus Carboplatin or Nab Paclitaxel Plus Carboplatin Versus Paclitaxel Plus Carboplatin Alone as First-Line Treatment for Untreated Advanced Squamous Non-small Cell Lung Cancer
Brief Title: A Study of Tislelizumab in Combination With Chemotherapy Versus Chemotherapy in Advanced Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-307; CTR20180292 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2018-07-03; First posted 2018-07-20 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tislelizumab + Paclitaxel + Carboplatin (Experimental): Tislelizumab 200 milligrams (mg) plus paclitaxel 175 mg/m^2 and carboplatin area under the plasma or serum concentration-time curve (AUC) 5 on Day 1 administered intravenously once every 3 weeks until unacceptable toxicity, withdrawal of consent, loss of clinical benefit, or disease progression; paclitaxel and carboplatin were administered for 4 to 6 cycles (each cycle is 21 days)
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Carboplatin
- Tislelizumab + Nab-paclitaxel + Carboplatin (Experimental): Tislelizumab 200 mg on Day 1 plus Nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 and carboplatin AUC 5 on Day 1 administered intravenously once every 3 weeks until unacceptable toxicity, withdrawal of consent, loss of clinical benefit, or disease progression; Nab-paclitaxel and carboplatin were administered for 4 to 6 cycles (each cycle is 21 days)
  Interventions: Drug: Tislelizumab; Drug: Nab-paclitaxel; Drug: Carboplatin
- Paclitaxel + Carboplatin (Active Comparator): Paclitaxel 175 mg/m^2 and carboplatin AUC 5 on Day 1 administered intravenously once every 3 weeks for 4 to 6 cycles (each cycle is 21 days)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously as described
  Other Names: BGB-A317; Tevimbra
  Arms: Tislelizumab + Nab-paclitaxel + Carboplatin; Tislelizumab + Paclitaxel + Carboplatin
Drug: Paclitaxel — Administered intravenously as described
  Arms: Paclitaxel + Carboplatin; Tislelizumab + Paclitaxel + Carboplatin
Drug: Nab-paclitaxel — Administered intravenously as described
  Arms: Tislelizumab + Nab-paclitaxel + Carboplatin
Drug: Carboplatin — Administered intravenously as described

SUMMARY:
An open-label, randomized, multicenter Phase 3 study designed to compare the efficacy and safety of tislelizumab combined with chemotherapy versus chemotherapy only as first-line treatment in advanced squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18-75 years old, male or female, and signed informed consent form (ICF)
2. Advanced NSCLC diagnosed by pathological or clinical physicians
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1
4. Participants must have ≥ 1 measurable lesion as defined per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
5. Must be treatment-naive for locally advanced or metastatic squamous NSCLC
6. Life expectancy ≥ 12 weeks
7. Participants must have adequate organ function
8. Male/Female is willing to use a highly effective method of birth control

Key Exclusion Criteria:

1. Diagnosed with NSCLC but with epidermal growth factor receptors (EGFR)-sensitizing mutation or anaplastic lymphoma kinase (ALK) gene translocation
2. Received any approved systemic anticancer therapy
3. Received prior treatment with EGFR inhibitors or ALK inhibitors
4. Received prior therapies targeting programmed death 1 (PD-1) or programmed death ligand 1 (PD-L1)
5. With history of interstitial lung disease
6. Clinically significant pericardial effusion
7. Severe infections, active leptomeningeal disease or uncontrolled, untreated brain metastasis
8. Any major surgical procedure before randomization
9. Human immunodeficiency virus infection
10. Untreated hepatitis B virus (HBV)/hepatitis C virus (HCV)
11. Active autoimmune diseases or history of autoimmune diseases
12. History of allergic reactions to chemotherapy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (43):
- China (43):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hangzhou First Peoples Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang J, Lu S, Yu X, Hu Y, Sun Y, Wang Z, Zhao J, Yu Y, Hu C, Yang K, Feng G, Ying K, Zhuang W, Zhou J, Wu J, Leaw SJ, Zhang J, Lin X, Liang L, Yang N. Tislelizumab Plus Chemotherapy vs Chemotherapy Alone as First-line Treatment for Advanced Squamous Non-Small-Cell Lung Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):709-717. doi: 10.1001/jamaoncol.2021.0366. PMID 33792623
- [Background] Wang, J, S. Lu, et al. Randomized Phase III Study of Tislelizumab plus Chemotherapy versus Chemotherapy Alone as First-Line Treatment for Advanced Squamous Non-Small Cell Lung Cancer (Sq-NSCLC): RATIONALE-307 Updated Analysis. IOTECH Abstract, Vol. 16 Supplement 1, Dec. 2022. doi.org/10.1016/j.iotech.2022.100244.
- [Derived] Duan J, Zhang Y, Chen R, Liang L, Huo Y, Lu S, Zhao J, Hu C, Sun Y, Yang K, Chen M, Yu Y, Ying J, Huang R, Ma X, Leaw S, Bai F, Shen Z, Cai S, Gao D, Wang J, Wang Z. Tumor-immune microenvironment and NRF2 associate with clinical efficacy of PD-1 blockade combined with chemotherapy in lung squamous cell carcinoma. Cell Rep Med. 2023 Dec 19;4(12):101302. doi: 10.1016/j.xcrm.2023.101302. Epub 2023 Dec 4. PMID 38052215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple study centers in China. Data are presented as of the study completion data cut-off date of 28APR2023.
Period: Overall Study
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Started | 120 | 119 | 121
Randomized But Not Treated | 0 | 1 | 4
Completed | 0 | 0 | 0
Not Completed | 120 | 119 | 121
Not completed — Death | 78 | 86 | 87
Not completed — Withdrawal by Subject | 5 | 2 | 11
Not completed — Lost to Follow-up | 4 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Sponsor decision | 23 | 17 | 16
Not completed — Did not meet inclusion criteria | 0 | 0 | 1
Not completed — Transfer to long term extension study | 10 | 12 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who were randomized. Data are presented as of the study completion data cut-off date of 28APR2023.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 120 | 119 | 121 | 360
Age, Continuous [Median (Full Range); unit: Years] | 60.0 [41 to 75] | 64.0 [38 to 74] | 63.0 [34 to 75] | 62.5 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 10 | 30
  Male | 107 | 112 | 111 | 330
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 120 | 119 | 121 | 360
  Not Hispanic or Latino | 120 | 119 | 121 | 360

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Independent Review Committee (IRC) Assessment as of Data Cut-off Date of 06DEC2019
Description: PFS is defined as the time from randomization until first documentation of disease progression as assessed by the IRC per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurs first
Time Frame: Through primary analysis data cut-off date of 06DEC2019 (up to approximately 1 year and 4 months)
Population: ITT analysis set included all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 119 | 121
Months | 7.6 [5.95 to 9.79] | 7.6 [5.75 to 11.01] | 5.5 [4.21 to 5.65]
Statistical Analysis 1: Comparison: Tislelizumab + Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.0001, One-sided stratified log-rank test; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.37 to 0.74]
Statistical Analysis 2: Comparison: Tislelizumab + Nab-paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority; p < 0.0001, One-sided stratified log-rank test; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.33 to 0.67]

2. Primary Outcome: PFS by IRC Assessment as of Data Cut-off Date of 30SEP2020
Description: PFS is defined as the time from randomization until first documentation of disease progression as assessed by the IRC per RECIST v1.1 or death from any cause, whichever occurs first
Time Frame: Through primary analysis data cut-off date of 30SEP2020 (up to approximately 2 years and 2 months)
Population: ITT analysis set included all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 119 | 121
Months | 7.7 [6.74 to 10.41] | 9.6 [7.39 to 10.78] | 5.5 [4.21 to 5.59]
Statistical Analysis 1: Comparison: Tislelizumab + Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.32 to 0.61]
Statistical Analysis 2: Comparison: Tislelizumab + Nab-paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.30 to 0.59]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until the date of death due to any cause
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 119 | 121
Months | 26.1 [18.99 to 33.81] | 23.3 [18.76 to 26.38] | 19.4 [15.97 to 23.43]

4. Secondary Outcome: Objective Response Rate (ORR) by IRC Assessment
Description: ORR is defined as the percentage of participants with complete response (CR) and partial response (PR), as assessed by the IRC using RECIST v1.1.
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 119 | 121
Percentage of participants | 74.2 [65.4 to 81.7] | 73.9 [65.1 to 81.6] | 47.9 [38.8 to 57.2]

5. Secondary Outcome: ORR by Investigator Assessment
Description: ORR is defined as the percentage of participants with complete response (CR) and partial response (PR), as assessed by the investigator using RECIST v1.1.
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 119 | 121
Percentage of participants | 70.0 [61.0 to 78.0] | 78.2 [69.6 to 85.2] | 49.6 [40.4 to 58.8]

6. Secondary Outcome: Duration of Response (DOR) by IRC Assessment
Description: DOR is defined as the time from the first occurrence of a documented objective response to the time of documented disease progression assessed by the IRC using RECIST v1.1, or death from any cause, whichever comes first, in all randomized participants with documented objective responses. Data are based on number of responders.
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 89 | 88 | 58
Months | 8.4 [5.03 to 18.69] | 8.6 [7.13 to 12.48] | 4.3 [2.86 to 5.42]

7. Secondary Outcome: DOR by Investigator Assessment
Description: DOR is defined as the time from the first occurrence of a documented objective response to the time of documented disease progression assessed by the investigator using RECIST v1.1, or death from any cause, whichever comes first, in all randomized participants with documented objective responses. Data are based on number of responders.
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 84 | 93 | 60
Months | 10.6 [7.03 to 16.23] | 8.8 [8.05 to 11.93] | 4.8 [2.86 to 6.11]

8. Secondary Outcome: PFS by Investigator Assessment
Description: PFS is defined as the time from randomization until first documentation of disease progression as assessed by the investigator per RECIST v1.1 or death from any cause, whichever occurs first
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 119 | 121
Months | 9.6 [7.62 to 11.76] | 9.8 [8.57 to 11.86] | 5.5 [4.17 to 5.65]

9. Secondary Outcome: PFS by IRC Based on Programmed Death Ligand 1 (PD-L1) Expression
Description: PFS is defined as the time from randomization until first documentation of disease progression as assessed by the IRC per RECIST v1.1 or death from any cause, whichever occurs first, based on PD-L1 expression in tumor cells
Time Frame: Through study completion data cut-off date of 28APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all participants who were randomized; participants evaluable for PD-L1 expression were included
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 119 | 118 | 117
Months
  PD-L Expression (<1%): number analyzed (Participants) | 47 | 46 | 45
  PD-L Expression (<1%) | 7.6 [5.5 to 14.5] | 7.6 [5.4 to 9.9] | 5.5 [4.2 to 7.0]
  PD-L Expression (1% to 49%): number analyzed (Participants) | 30 | 30 | 31
  PD-L Expression (1% to 49%) | 9.9 [5.5 to 22.7] | 9.8 [7.6 to 12.0] | 5.0 [2.8 to 6.5]
  PD-L Expression (≥ 50%): number analyzed (Participants) | 42 | 42 | 41
  PD-L Expression (≥ 50%) | 7.7 [5.9 to 9.8] | 9.7 [5.6 to 30.9] | 5.5 [4.1 to 5.6]

10. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer (EORTC QLQ-LC13)
Description: Least squares mean change from baseline in EORTC QLQ-CL13 scores for chest pain, coughing, and dyspnea between tislelizumab arms and paclitaxel + carboplatin arm. The EORTC QLQ-LC13 is a questionnaire that measures lung cancer-specific disease and treatment symptoms. It includes questions about specific symptoms in which participants respond based on a 4-point scale, where 1 is "not at all" and 4 is "very much". Raw scores are transformed into a 0 to 100 scale via linear transformation. A lower score indicates an improvement in symptoms.
Time Frame: Baseline to Cycle 5; each cycle is 21 days
Population: Health-Related Quality of Life (HRQoL) analysis set included all randomized participants who received ≥ 1 dose of study drug and completed ≥ HRQoL assessment post baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 118
Score on a scale
  Chest pain | 0.4 [-5.0 to 5.9] | -0.4 [-5.9 to 5.1]
  Coughing | -7.0 [-14.3 to 0.2] | -0.4 [-7.7 to 6.8]
  Dyspnea | -2.7 [-6.9 to 1.6] | -1.0 [-5.3 to 3.3]

11. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status
Description: Least squares mean change from baseline in EORTC QLQ-C30 Global Health Status/Quality of Life score between tislelizumab arms and paclitaxel + carboplatin arm. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of cancer patients. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 5; each cycle is 21 days
Population: HRQoL analysis set included all randomized participants who received ≥ 1 dose of study drug and completed ≥ HRQoL assessment post baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 118
Score on a scale | 2.4 [-3.4 to 8.2] | 3.3 [-2.5 to 9.2]

12. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), which includes laboratory tests, physical exams, electrocardiogram results and vital signs, according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Time Frame: From first dose to 30 days after the last dose (up to approximately 4 years and 9 months)
Population: Safety analysis set included all randomized participants who received ≥ 1 dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 120 | 118 | 117
Participants
  At least 1 TEAE | 120 | 117 | 117
  At least 1 SAE | 56 | 55 | 29

ADVERSE EVENTS:
Time Frame: From the first dose up to 30 days after the last dose of study drug, up to approximately 4 years and 9 months
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events includes all randomized participants who received ≥ 1 dose of any study treatment
Arm/Group | Tislelizumab + Paclitaxel + Carboplatin | Tislelizumab + Nab-Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 78/120 | 86/119 | 87/121
Serious Adverse Events (participants affected / at risk) | 56/120 | 55/118 | 29/117
Other Adverse Events (participants affected / at risk) | 119/120 | 117/118 | 116/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Paclitaxel + Carboplatin (N=120) | Tislelizumab + Nab-Paclitaxel + Carboplatin (N=118) | Paclitaxel + Carboplatin (N=117)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 12 (15) | 7 (7) | 5 (5)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cerebral radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram ST-T segment abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 4 (5) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Paclitaxel + Carboplatin (N=120) | Tislelizumab + Nab-Paclitaxel + Carboplatin (N=118) | Paclitaxel + Carboplatin (N=117)
Anaemia (Blood and lymphatic system disorders) | 107 (277) | 111 (297) | 94 (198)
Leukocytosis (Blood and lymphatic system disorders) | 3 (4) | 4 (5) | 7 (11)
Leukopenia (Blood and lymphatic system disorders) | 58 (234) | 66 (291) | 57 (187)
Neutropenia (Blood and lymphatic system disorders) | 53 (191) | 50 (196) | 56 (160)
Thrombocytopenia (Blood and lymphatic system disorders) | 36 (89) | 48 (131) | 33 (54)
Sinus bradycardia (Cardiac disorders) | 2 (6) | 5 (12) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 4 (4) | 5 (14) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 6 (6) | 1 (7) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 7 (9) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 19 (42) | 16 (26) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 10 (12) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 7 (10) | 7 (8) | 3 (3)
Constipation (Gastrointestinal disorders) | 40 (48) | 36 (50) | 27 (30)
Diarrhoea (Gastrointestinal disorders) | 21 (32) | 24 (41) | 8 (9)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 5 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 37 (68) | 54 (87) | 35 (51)
Oral pain (Gastrointestinal disorders) | 2 (2) | 4 (6) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 4 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 28 (41) | 26 (41) | 19 (25)
Asthenia (General disorders) | 30 (38) | 24 (32) | 23 (33)
Chest discomfort (General disorders) | 5 (5) | 5 (6) | 1 (1)
Chest pain (General disorders) | 5 (6) | 4 (4) | 3 (3)
Fatigue (General disorders) | 5 (8) | 6 (6) | 6 (6)
Malaise (General disorders) | 22 (35) | 19 (32) | 19 (31)
Non-cardiac chest pain (General disorders) | 5 (5) | 5 (7) | 2 (2)
Oedema peripheral (General disorders) | 3 (5) | 7 (12) | 2 (2)
Pain (General disorders) | 8 (10) | 3 (3) | 6 (10)
Pyrexia (General disorders) | 25 (32) | 24 (40) | 17 (23)
Hepatic function abnormal (Hepatobiliary disorders) | 7 (11) | 3 (3) | 10 (11)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 3 (4) | 4 (5)
Influenza (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 15 (25) | 13 (17) | 8 (10)
Rash pustular (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 20 (25) | 15 (23) | 11 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (6) | 5 (8) | 4 (7)
Alanine aminotransferase increased (Investigations) | 57 (131) | 46 (82) | 27 (42)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 6 (10) | 2 (5) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 52 (120) | 44 (82) | 14 (19)
Bilirubin conjugated increased (Investigations) | 6 (9) | 4 (9) | 4 (5)
Blood albumin decreased (Investigations) | 2 (2) | 5 (9) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 20 (33) | 12 (21) | 11 (18)
Blood bilirubin increased (Investigations) | 31 (94) | 21 (46) | 15 (22)
Blood bilirubin unconjugated increased (Investigations) | 5 (9) | 5 (10) | 4 (6)
Blood chloride decreased (Investigations) | 6 (6) | 2 (3) | 2 (3)
Blood cholesterol increased (Investigations) | 3 (13) | 2 (2) | 4 (5)
Blood creatine phosphokinase MB increased (Investigations) | 5 (10) | 6 (12) | 1 (2)
Blood creatine phosphokinase decreased (Investigations) | 4 (6) | 2 (3) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 22 (47) | 16 (56) | 10 (14)
Blood creatinine increased (Investigations) | 7 (12) | 11 (36) | 7 (10)
Blood fibrinogen increased (Investigations) | 3 (3) | 4 (14) | 2 (3)
Blood glucose increased (Investigations) | 6 (8) | 2 (2) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 23 (45) | 20 (33) | 13 (20)
Blood magnesium decreased (Investigations) | 4 (6) | 2 (2) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1) | 5 (5) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 4 (4) | 9 (17) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 10 (15) | 9 (24) | 1 (1)
Blood urea increased (Investigations) | 7 (9) | 4 (5) | 4 (7)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 5 (7) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 4 (6) | 4 (20) | 0 (0)
Fibrin D dimer increased (Investigations) | 4 (4) | 4 (10) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 21 (47) | 18 (30) | 15 (20)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 5 (9) | 0 (0)
Lymphocyte count decreased (Investigations) | 16 (38) | 24 (84) | 16 (32)
Neutrophil count decreased (Investigations) | 78 (283) | 73 (327) | 68 (220)
Neutrophil count increased (Investigations) | 6 (7) | 5 (5) | 2 (2)
Platelet count decreased (Investigations) | 45 (109) | 54 (137) | 29 (64)
Protein total decreased (Investigations) | 1 (1) | 2 (13) | 5 (7)
Thyroxine free decreased (Investigations) | 2 (2) | 6 (9) | 1 (1)
Thyroxine free increased (Investigations) | 0 (0) | 6 (12) | 0 (0)
Total bile acids increased (Investigations) | 5 (6) | 5 (7) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 3 (3) | 4 (5) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 1 (1) | 7 (8) | 0 (0)
Urinary occult blood positive (Investigations) | 1 (1) | 4 (5) | 0 (0)
Weight decreased (Investigations) | 15 (18) | 17 (22) | 8 (8)
Weight increased (Investigations) | 13 (17) | 9 (15) | 2 (2)
White blood cell count decreased (Investigations) | 68 (241) | 68 (291) | 61 (190)
White blood cell count increased (Investigations) | 4 (4) | 5 (5) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 55 (87) | 55 (89) | 37 (72)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (10) | 3 (3) | 4 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 (19) | 7 (12) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 22 (65) | 15 (34) | 10 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (7) | 4 (5)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 4 (5) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 (30) | 8 (27) | 8 (12)
Hyperuricaemia (Metabolism and nutrition disorders) | 18 (50) | 15 (71) | 6 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 32 (56) | 27 (40) | 19 (26)
Hypocalcaemia (Metabolism and nutrition disorders) | 15 (23) | 10 (31) | 5 (7)
Hypochloraemia (Metabolism and nutrition disorders) | 11 (19) | 11 (17) | 11 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 27 (42) | 22 (40) | 16 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (13) | 9 (16) | 7 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 28 (47) | 28 (59) | 20 (29)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (9) | 7 (20) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 17 (33) | 11 (23) | 12 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (61) | 29 (38) | 20 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (17) | 20 (22) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 6 (10)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (7) | 6 (8) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (9) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (9) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 (59) | 20 (35) | 27 (38)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 4 (6) | 6 (6)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 6 (8) | 10 (11) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 6 (7) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 27 (35) | 13 (13) | 20 (30)
Neurotoxicity (Nervous system disorders) | 15 (16) | 6 (6) | 12 (14)
Paraesthesia (Nervous system disorders) | 5 (7) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (10) | 1 (1) | 5 (6)
Insomnia (Psychiatric disorders) | 9 (14) | 11 (13) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 19 (22) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 15 (17) | 11 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 17 (23) | 13 (18)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 10 (10)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 78 (80) | 82 (84) | 72 (73)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 9 (10) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 25 (36) | 28 (31) | 4 (5)
Hypertension (Vascular disorders) | 5 (5) | 6 (10) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03594747/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT03594747/SAP_001.pdf